CLINICAL TRIAL: NCT03335241
Title: An Open-label, Randomised Phase II Study of Fludarabine With Pegylated Liposomal Doxorubicin Versus Pegylated Liposomal Doxorubicin Alone In Patients With Platinum Resistant/Refractory Ovarian Cancer
Brief Title: Study of Fludarabine With Pegylated Liposomal Doxorubicin Versus Pegylated Liposomal Doxorubicin Alone In Patients With Platinum Resistant/Refractory Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jundong Li, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 308-2016-03-01
Record Dates: First submitted 2017-11-01; First posted 2017-11-07 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Fludarabine; Pegylated Liposomal Doxorubicin; Chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — fludarabine; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Fludarabine and Pegylated liposomal doxorubicin (Experimental)
  Interventions: Drug: Fludarabine and Pegylated liposomal doxorubicin
- Arm 2: Pegylated liposomal doxorubicin (Active Comparator)
  Interventions: Drug: Pegylated liposomal doxorubicin

INTERVENTIONS:
Drug: Fludarabine and Pegylated liposomal doxorubicin — Fludarabine 25mg/m2 iv on days d1-d3 of each 4-week cycle
  Pegylated liposomal doxorubicin 30mg/m2 iv every 4 weeks
  Arms: Arm 1: Fludarabine and Pegylated liposomal doxorubicin
Drug: Pegylated liposomal doxorubicin — Pegylated liposomal doxorubicin 50mg/m2 iv every 4 weeks
  Arms: Arm 2: Pegylated liposomal doxorubicin

SUMMARY:
The purpose of the study is to evaluate the efficacy and toxicity of fludarabine with pegylated liposomal doxorubicin versus pegylated liposomal doxorubicin alone in patients with platinum resistant or refractory ovarian cancer.

DETAILED DESCRIPTION:
Ovarian cancer is the leading cause of death for patients with gynecologic malignancies. Approximately 75% of patients are diagnosed at an advanced stage will eventually experience disease recurrence. The overall response rates of second-line chemotherapy for recurrent ovarian cancer are only 20-27%. The 5-year overall survival rates are less than 20%. Therefore, it is important to seek alternative agent that can improve the outcome. Fludarabine is a purine nucleoside analog prodrug that upon phosphorylation is toxic to dividing and quiescent lymphocytes and monocytes, exerting its effects through DNA synthesis interference and apoptosis. The preclinical studies suggest fludarabine may be effective in other cancers such as ovarian cancer. Therefore, the purpose of this study is to test the efficacy and safety of the study drug fludarabine combined with pegylated liposomal doxorubicin versus pegylated liposomal doxorubicin alone in patients with platinum resistant or refractory ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or pathologically confirmed diagnosis of epithelial carcinoma of the ovary.
* Platinum resistant or refractory ovarian cancer
* At least treated with one line of platinum-based chemotherapy
* Female, age ≥18 years and ≤70 years, signed informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 version
* Patients must have a life expectancy of at least 3 months.
* Patients must have adequate organ function as defined by the following criteria:

  * White blood cell count ≥ 3 x 10^9/L, Absolute neutrophil count (ANC) (≥ 1.0 x 10^9/L), Hemoglobin of ≥ 80 g/L, Platelets ≥ 80 x 10^9/L
  * Total bilirubin ≤ 1 x upper limit of normal (ULN), AST and ALT ≤ 2.5 x ULN
  * Serum creatinine ≤ 1 x ULN
* Symptomatic central nervous system (CNS) metastasis

Exclusion Critera:

* Has known allergies to any of the excipients.
* Prior treatment with adriamycin or other anthracycline at cumulative doses greater than 550 mg/m2 after 6 cycles of pegylated liposomal doxorubicin
* LVEF (left ventricular ejection fraction) <50%
* Had disease recurrence/progression within 6 months after the administration of doxorubicin chemotherapy
* History of myocardial infarction, or unstable angina, or New York Heart Association (NYHA) Grade III-IV within 6 months prior to Day 1.
* Known significant chronic liver disease, such as cirrhosis or active hepatitis
* Uncontrollable active infection

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to four years
  Progression-free survival estimated using Kaplan-Meier methods is defined as the time from registration to the earlier of death or disease progression. Patients alive without disease progression are censored at the date of last disease evaluation. Progressive disease (PD) based on RECIST 1.0 is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Equivocal progression of non-target lesions also qualifies as PD

SECONDARY OUTCOMES:
Objective response rate | Up to four years
  Objective response rate defined as confirmed complete response or partial response under RECIST 1.0 criteria. CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. To be assigned a status of CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed no fewer than 4 weeks after the response criteria are first met.

OTHER OUTCOMES:
Frequency and severity of adverse effects as defined by CTCAE version 4.0 | 30 days after last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes